CLINICAL TRIAL: NCT05732194
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ITI-333 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ITI 333 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ITI-333-002; 1UG3DA047699-02 (NIH); 1UG3DA047699 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Sequential ascending doses. Parallel (active, placebo) within each cohort
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: 0.75 mg ITI-333 or placebo once daily for 14 days (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 2: 1.5 mg ITI-333 or placebo once daily for 14 days (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 3: 3 mg ITI-333 or placebo once daily for 14 days (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo
- Cohort 4: 6 mg ITI-333 or placebo once daily for 14 days (Experimental)
  Interventions: Drug: ITI-333; Other: Placebo

INTERVENTIONS:
Drug: ITI-333 — ITI-333 oral solution
Other: Placebo — Matching placebo

SUMMARY:
The study will be conducted as a single-center, randomized, double-blind, placebo-controlled, ascending dose study in up to 4 sequential cohorts of healthy subjects. Each cohort will enroll 8 subjects: 6 subjects will receive ITI-333 and 2 subjects will receive placebo once daily for 14 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female subjects between 18 and 45 years old (inclusive);
* BMI inclusive of 18-32 kg/m2 at screening and a minimum weight of 50 kg;
* Willingness to remain in the clinic for the inpatient portion of the study and return for follow-up visit(s) as required by protocol and as deemed necessary by the Investigator.

Key Exclusion Criteria:

* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the subject at risk or interfere with study outcome variables; this includes, but is not limited to, history of or current cardiac, hepatic, renal, neurologic, GI, pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy;
* Clinically significant abnormal findings in vital sign assessments, including blood oxygen saturation (SpO2) < 96% and respiratory rate < 12 breaths per min;
* History of psychiatric condition that in the Investigator's opinion may be detrimental to participation in the study;
* CRP, ESR, or fibrinogen that are above normal reference ranges at Screening or Day 1.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: AUC0-tau | Day 14
  Area under the plasma drug concentration-time curve (AUC) from time zero to the end of dosing interval
Pharmacokinetics: Cmax | Day 14
  Maximum plasma concentration of ITI-333 over a dosing interval
Pharmacokinetics: Tmax | Day 14
  Time of maximum plasma concentration of ITI-333 over a dosing interval
Percentage of subjects with treatment-emergent adverse events | up to 30 days after last dose
Change from baseline in systolic and diastolic blood pressure | Baseline and Day 17
Change from baseline in SpO2 | Baseline and Day 17
Change from baseline in ECG QT interval | Baseline and Day 17
Change from baseline in aspartate aminotransferase | Baseline and Day 17
Change from baseline in alanine aminotransferase | Baseline and Day 17

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site 1, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No